CLINICAL TRIAL: NCT06069063
Title: Double Blind Placebo-controlled Crossover Study of Zafirlukast in Preventing Allergen-induced Signs and Symptoms of Allergic Rhinitis in Response to Cat Dander Challenge
Brief Title: Crossover Study of Zafirlukast in Preventing Allergen-induced Signs and Symptoms in Response to Cat Dander Challenge
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Allergy & Asthma Medical Group & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACC001
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Allergy to Cats
MeSH Terms: interventions — zafirlukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zafirlukast cross-over to Placebo (Experimental): This group will receive the Zafirlukast pre-treatment nasally (400 mcg in 150 mcl in each nostril) once before the allergen challenge (0.87mcg Fel d1 in 100mcl in each nostril) in the first study visit. In the second study visit, they will receive a placebo pre-treatment nasally (150 mcl each nostril) once before the allergen challenge (0.87mcg Fel d1 in 100mcl in each nostril).
  Interventions: Drug: Zafirlukast
- Placebo cross-over to Zafirlukast (Experimental): This group will receive a placebo pre-treatment nasally (150 mcl each nostril) once before the allergen challenge (0.87mcg Fel d1 in 100mcl in each nostril) in the first study visit. In the second study visit, they will receive the Zafirlukast pre-treatment nasally (400 mcg in 150 mcl in each nostril) once before the allergen challenge (0.87mcg Fel d1 in 100mcl in each nostril).
  Interventions: Drug: Zafirlukast

INTERVENTIONS:
Drug: Zafirlukast — Oral zafirlukast is approved to treat asthma and been shown in previous trials to be effective in blocking or mitigating the symptoms of people allergic to cat dander

SUMMARY:
The goal of this clinical trial is to test the hypothesis that pre-treatment with a nasal dose of Zafirlukast works well in blocking the signs and symptoms of cat dander in patients sensitive to cat dander. The main question it aims to answer is:

• What is the difference in the symptoms of patients pre-treated with Zafirlukast and patients treated with a placebo (a look-alike substance that contains no active drug) when exposed to cat dander?

Participants will screened to see if they qualify for the study based on their reaction to being exposed to cat dander and medical history. If they qualify, they will make two more visits to the allergy center, where they will be pre-treated with either Zafirlukast or a placebo and exposed to cat dander, then observed for four hours.

Participants will

* First be screened for their medical history, the medication they take, and other factors to see if they qualify for the study.

  * Participants will then be exposed to a fixed dose of cat dander to test their baseline change in TNSS. Some patients may need to return for a higher dose of cat dander.
* On the next visit, some participants will be pre-treated with Zafirlukast and the rest with a placebo, then they will be exposed to cat dander. Their symptoms will be observed.
* On the final visit, participants who were pre-treated with Zafirlukast on their last visit will be given a placebo. Participants who were pre-treated with a placebo on their last visit will be given Zafirlukast. All participants will then be exposed to cat dander and their symptoms will be observed.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test the hypothesis that pre-treatment with a nasal dose of Zafirlukast works well in blocking the signs and symptoms of cat dander in patients sensitive to cat dander. The main question it aims to answer is:

• What is the difference in the Total Nasal Symptoms Score between patients pre-treated with Zafirlukast and patients treated with a placebo (a look-alike substance that contains no active drug)?

The Total Nasal Symptom Score (TNSS; possible score of 0-12) is the sum of 4 individual subject-assessed symptom scores for

* rhinorrhea (runny nose)
* nasal congestion (stuffy nose)
* nasal itching
* sneezing

Each of these are evaluated using a scale of

* 0=None
* 1=Mild
* 2=Moderate
* 3=Severe

Participants will

* First be screened for their medical history, the medication they take, and other factors to see if they qualify for the study.
* Participants will then be exposed to a fixed dose of cat dander to test their baseline change in TNSS. Some patients may need to return for a higher dose of cat dander.
* On the next visit, some participants will be pre-treated with Zafirlukast and the rest with a placebo, then they will be exposed to cat dander. Their symptoms will be observed.
* On the final visit, participants who were pre-treated with Zafirlukast on their last visit will be given a placebo. Participants who were pre-treated with a placebo on their last visit will be given Zafirlukast. All participants will then be exposed to cat dander and their symptoms will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Active nonsmoking males and females between the ages of 18-65 with allergic rhinitis triggered by cat dander exposure.
* Concomitant medication limited to "as needed" including for mild asthma.
* Baseline resting blood pressure les than or equal to 140/90 mm Hg.
* Baseline resting heart rate less than or equal to 100 beats/min.
* Baseline NIFR must be ≥ 50 L/min.
* Females of childbearing age may participate only if they have a negative urine pregnancy test, are non-lactating, and agree to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for the duration of the study.
* The ability to give informed consent and comply with study procedures.

Exclusion Criteria:

* Receiving immunotherapy for cat allergy
* Predictable seasonal allergy during the study period
* Newly (< 2 weeks) diagnosed with Corona Virus Disease (COVID-19)
* Regular use of controller medication for moderate to severe asthma
* Subject works with cats or keeps a cat as a pet.
* Inability or unwillingness to give written informed consent.
* History of upper/lower respiratory tract infection, requiring systemic steroids, antibiotics, and or emergency room (ER) visit or urgent care within 6 weeks of screening visit.
* History of adverse reaction or allergy to Zafirlukast
* History of neurological, hepatic, renal, diabetic mellitus, thyroid disorder, psychiatric, addiction or other medical conditions that may interfere with the interpretation of data or the patient's participation in the study or may increase safety concerns per investigator discretion.
* History of cardiovascular diseases including uncontrolled hypertension (blood pressure >160/100 mmHg), ischemic heart disease, congestive heart failure (New York Heart Association III or IV), valvular heart disease or cardiomyopathy (e.g., depressed left ventricular ejection fraction by echo, arrhythmias).
* Known allergy or sensitivity to atropine or ipratropium bromide.
* Documented or self-reported current history of alcoholism or drug abuse.
* Baseline Spirometry Forced Expiratory Volume in first second (FEV1) <70% of predicted
* Participated in another research trial and received investigational drug within 30 days or 5 half-lives, whichever is longer
* Unwillingness or inability to comply with study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | Starts at 10 minutes after the cat allergen challenge, then 30, 60, 120, and 240 minutes after.
  The Total Nasal Symptom Score (TNSS; possible score of 0-12) is the sum of 4 individual subject-assessed symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe.

SECONDARY OUTCOMES:
Total Ocular Symptom Score (TOSS) | Starts at 10 minutes after the cat allergen challenge, then 30, 60, 120, and 240 minutes after.
  The Total Ocular Symptom Score (TOSS; possible score of 0-12) is the sum of 4 individual subject-assessed symptom scores for itchiness, redness, tearing, and swelling, each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe.
Nasal Inspiratory Flow Rate (NIFR) | Starts at 10 minutes after the cat allergen challenge, then 30, 60, 120, and 240 minutes after.
  NIFR is an inexpensive, rapid, easy-to-use objective measure that directly measures nasal airflow during maximal inspiration. NIFR is measured in L/min.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Greiner, MD, Principal Investigator — Allergy & Asthma Medical Group & Research Center

IPD SHARING:
Plan to Share IPD: No